CLINICAL TRIAL: NCT01876004
Title: Effectiveness Of Expectant Management In The Tubal Ectopic Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Priscila Matthiesen e Silva, Obstetrics and Gynecologist, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP UNIFESP 0772/11
Record Dates: First submitted 2013-06-06; First posted 2013-06-12 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Ectopic Pregnancy
Keywords: ectopic pregnancy; methotrexate; human chorionic gonadotropin beta subunit; expectant management
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate (Experimental): Administered a single intramuscular dose of 50 mg/m2 of Methotrexate.
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Prescribed Placebo intramuscularly.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — 50 mg/m2, IM (intramuscularly), single dose
  Arms: Methotrexate
Drug: Placebo — Prescribed Placebo IM (intramuscularly), single dose
  Arms: Placebo

SUMMARY:
Objectives: To evaluate if, when considering expectant management in tubal ectopic pregnancy if the complementary use of Methotrexate could provide better results. We evaluate the success of treatment and the time required for titers of β-hCG to become negative. Methods: A double-blind randomized study, held at the Department of Obstetrics UNIFESP. The patients will be divided into two groups: in one patients will be administered a single intramuscular dose of 50 mg/m2 of Methotrexate and in the other patients will be prescribed Placebo intramuscularly. The monitoring will be done by measurement of β-hCG in the 4th and 7th day. When the decline of beta-hCG titers was > 15% in this interval, the patient was followed with weekly dosing of β-hCG until the titers become negative. The criterion of success is when the β-hCG was negative. The treatment failure occurs when surgery was necessary.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamic stability
* Initial β-hCG <2000 mIU / mL
* Titers of β-hCG in decline in 48 hours before treatment
* Adnexal mass <5.0 cm
* Desire for future pregnancy

Exclusion Criteria:

* Alive embryo
* Ectopic pregnancy other than in tubal location
* Pregnancy of unknown location

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
success of treatment | 6 months
  β-hCG negative (<5 mIU / mL)
Time required for titers of β-hCG to become negative | 6 weeks
  After medication, monitoring will be done by measurement of β-hCG in the 4th and 7th day. If there ia a decrease > 15% in this range (4th and 7th), patient will be followed with weekly dosing of β-hCG until negative titers

SECONDARY OUTCOMES:
Blood tests before treatment with Methotrexate and Placebo | 6 months
  Average value for tests: complete blood count, liver and renal function in the groups Methotrexate and Placebo before and after treatment
Blood tests after treatment with Methotrexate and Placebo | 6 months
  Average value for tests: complete blood count, liver and renal function in the groups Methotrexate and Placebo before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Julio Elito Junior, Study Director — Federal University of São Paulo; Luiz Camano, Study Director — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil